CLINICAL TRIAL: NCT04877080
Title: Exploratory Study to Evaluate Efficacy and Safety of Fast Dual CAR-T Injection in CD19+ Refractory or Relapsed B Cell Non-Hodgkinlymphoma
Brief Title: CD19 and BCMA Targeted Fast Dual CAR-T for CD19+ Refractory/Relapsed B-NHL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The PI decides to withdraw the research.
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 211
Record Dates: First submitted 2021-04-13; First posted 2021-05-07 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: B-cell Lymphoma
Keywords: Fast; CAR-T; CD19; B-NHL
MeSH Terms: conditions — Lymphoma, B-Cell; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fast Dual CAR-T treatment (Experimental): CD19+ R/R B-NHL patients be treated with a single dose of Fast Dual CAR-T cells. Total dose of (1-5)*10E5/kg cells will be administered at Day 0.
  Interventions: Biological: Fast Dual CAR-T Injection

INTERVENTIONS:
Biological: Fast Dual CAR-T Injection — Fast Dual CAR-T injection is a autologous dual CAR-T targeted CD19 and BCMA. A single infusion of CART cells will be administered intravenously.

SUMMARY:
This is a single arm, open-label, single-center prospective study to determine the safety and efficacy of Fast Dual CAR-T cells in patients diagnosed with CD19+ refractory/relapsed B cell non-Hodgkinlymphoma (R/R B-NHL).

DETAILED DESCRIPTION:
The main aim of the study is to determine the safety and efficacy of Fast Dual CAR-T in R/R B-NHL. Fast Dual CAR-T is an autologous dual chimeric antigen receptor T-cell (CAR-T) therapy that targets CD19 and B-cell maturation antigen (BCMA). The study will include 15 subjects to receive Fast Dual CAR-T single infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed: Diffuse Large B Cell Lymphoma (DLBCL), Transformation Follicular Lymphoma (TFL), Primary Mediastinal Large B Cell Lymphoma (PMBCL) and Mantle Cell Lymphoma (MCL), High-Grade B Cell Lymphoma (HGBL);

   1. Refractory B-NHL: PD as the best response to normative first-line therapy (intolerance of first-line therapy is not included in this study) or SD as the best response to at least 4 courses of first-line therapy with duration no longer than 6 month from last therapy; or PD as the best response to the last therapy of second-line therapy and above,or SD as the best response to at least 2 courses of second-line therapy with duration no longer than 6 month from last therapy, or:
   2. Relapsed B-NHL: Histopathology confirmed relapse after standard systemic and second-line therapy achieved CR, or histopathologically confirmed relapse within 1 year after autologous hematopoietic stem cell transplantation (Not limited by previous therapy);
   3. Prior therapy must include anti-CD20 monoclonal antibody (unless investigator determines that tumor is CD20-negative) and an anthracycline;
   4. For individual with TFL, must have chemotherapy and the conform the above definition of relapse or refractory after transformation;
2. According to the 2014 Lugano therapy response standard, there should be at least one measurable tumor focus: the longest diameter of nodular lesions> 1.5 cm, and the longest diameter of extranodal lesions> 1.0 cm;
3. CD19 positive expression in tumor tissue biopsy;
4. Prior to apheresis, approved anti-B-NHL therapys such as systemic chemotherapy, systemic radiotherapy and immunotherapy have been completed for at least 2 weeks;
5. Eastern cooperative oncology group (ECOG) performance status of 0 to 1;
6. Life expectancy ≥12 weeks;
7. Absolute neutrophil count (ANC)≥ 1×10^9/L;
8. Platelet count≥50×10^9/L;
9. Absolute lymphocyte count (ALC)≥1×10^8/L;
10. Adequate organ function defined as:

    1. Serum ALT/AST ≤2.5 ULN;
    2. Creatinine clearance (as estimated by Cockcroft Gault) ≥60 mL/min;
    3. PT and APTT≤1.5 ULN
    4. Total bilirubin ≤1.5 ULN;
    5. Cardiac ejection fraction ≥50%, no pericardial effusion, no clinically significant ECG findings;
    6. Baseline oxygen saturation >92% on room air;
11. Sufficient venous access for leukapheresis collection, and no other contraindications to leukapheresis;
12. Female of childbearing age must agree to take effective contraceptive measures at least 1 year after infusion; Male with fertile partners must agree to use effective barrier contraceptive methods at least 1 year after infusion;
13. Understand and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Diagnosis of other malignancy (except for cured non-melanoma skin cancer, cervical carcinoma in situ, superficial bladder cancer, ductal carcinoma in situ, or other malignancies that have completely responsed for more than 5 years);
2. Severe mental disorders;
3. History of hereditary diseases, including but not limited to: Fanconi anemia, Shut-Dai syndrome, Costman syndrome or any other known bone marrow failure syndrome;
4. History of allogeneic stem cell transplantation;
5. Grade III-IV heart failure or myocardial infarction, angioplasty or stent placement, unstableangina pectoris, or other clinically prominent heart disease within one year before enrollment.
6. Have any indwelling catheter or drainage tube (such as percutaneous nephrostomy tube, indwelling catheter, bile drainage tube or pleura / peritoneum / pericardial catheter), the use of dedicated central venous catheter is allowed;
7. Subjects with CNS lymphoma, cerebrospinal fluid malignant cells or brain metastases;
8. History or presence of CNS disorder, including but not limited to: seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement;
9. Positive for any of the following etiological tests: HIV, HBV, HCV, TPPA;
10. Presence of fungal, bacterial, viral, or other infection that is uncontrolled;
11. Allergic subjects or subjects with severe allergic reactions to cyclophosphamide or fludarabine;
12. History of autoimmune disease resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years;
13. History or diagnosis of pulmonary fibrosis;
14. Have received gene therapy or any other CAR-T treatment;
15. Have received any other drugs targeting CD19;
16. Subjects who received other clinical trial therapy within 4 weeks before participating in this trial, or the informed consent form was signed within the 5 half-life of the last administration in the other clinical trial (take longer time as standard);
17. Poor adherence due to physical, family, social, geographic, and other factors, who cannot follow the research plan and follow-up plan;
18. Subjects with comorbidities that require systemic corticosteroid therapy (≥5 mg/day of prednisone or an equivalent dose of other corticosteroids) or other immunosuppressive drugs within 6 months after study therapy according to the discretion of investigator;
19. Lactating women who are reluctant to stop breastfeeding;
20. Any other conditions defined by researcher that is inappropriate for the subject to be enrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-05 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE after Fast Dual CAR-T infusion | up to 24 weeks after Fast Dual CAR-T infusion
  Incidence of adverse events after Fast Dual CAR-T infusion

SECONDARY OUTCOMES:
ORR rate | 12 weeks, 24 weeks after Fast Dual CAR-T infusion
  Overall response rate (ORR=CR+CRi) after Fast Dual CAR-T infusion
PFS | 12 weeks, 24 weeks after Fast Dual CAR-T infusion
  Progression free survival (PFS) after Fast Dual CAR-T infusion
OS | 12 weeks, 24 weeks after Fast Dual CAR-T infusion
  overall survival (OS) after Fast Dual CAR-T infusion
Change of CAR Copies | Days 4, 7, 10, 14 and weeks 4, 8, 12, 18, 24 after Fast Dual CAR-T infusion
  CAR Copies measured by qPCR after Fast Dual CAR-T infusion
Change of CAR-T cell counts | Days 4, 7, 10, 14 and weeks 4, 8, 12, 18, 24 after Fast Dual CAR-T infusion
  CAR-T cell counts measured by Flow cytometry after Fast Dual CAR-T infusion
Changes in the concentration of cytokine IL-1, IL-2, IL-6, IL-10, TNF-α and IFN-γ. | Days 4, 7, 10, 14 and 28 after Fast Dual CAR-T infusion
  Cytokines in serum measured by ELISA after Fast Dual CAR-T infusion
Change of RCL in blood | Weeks 4, 12, 24 after Fast Dual CAR-T infusion
  Replication competent lentivirus (RCL) in blood after Fast Dual CAR-T infusion

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, Doctor, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China